CLINICAL TRIAL: NCT05840562
Title: Capsaicin 179 mg Patch Versus Oral Duloxetine in Patients With Chemotherapy-induced Peripheral Neuropathy : a Phase 3 Randomized Multicentric Open-label Study.
Brief Title: Capsaicin 179 mg Patch Versus Oral Duloxetine in Patients With Chemotherapy-induced Peripheral Neuropathy
Acronym: CAPNEUCHIM
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Institut Cancerologie de l'Ouest (Other)
Collaborators: Grünenthal GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ICO-2022-02
Record Dates: First submitted 2023-04-21; First posted 2023-05-03 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-08

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy
MeSH Terms: interventions — Capsaicin; Duloxetine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Arm (Experimental): The capsaicin 179 mg patch should be applied to the most painful extremities.
  Application:
  * Capsaicin patches must be applied to intact, dry and non-irritated skin and allowed to remain in place for 30 minutes for the feet and maximum 60 minutes for hands depending on immediate tolerance.
  * If all the areas to be treated cannot be treated in once, a second session will be organised between 3 and 7 days later. Further sessions can be held within 15 days of the 1st session (up to 4 sessions in total). All sessions will be considered as one application.
  * 1 application may require several treatment sessions.
  * The patch, which may be cut to shape, was used within 2 h of opening the foil pouch.
  After the first treatment session, treatment may be repeated every 2 months (at weeks 9, 17, 25) as warranted by the persistence or return of pain.
  Interventions: Drug: Capsaicin
- Control Arm (Active Comparator): Duloxetine should be initiated at an initial dose of 30 mg orally for 1 week followed by a maintenance dose of 60 mg per day, given either once a day or 30 mg orally 2 times a day.
  After W6, in case of insufficient response to the 60 mg dose, the dosage may be increased to the maximum dose of 120 mg.
  Interventions: Drug: Duloxetine

INTERVENTIONS:
Drug: Capsaicin — Application of capsaicin patches 179 mg
  Other Names: Qutenza
  Arms: Experimental Arm
Drug: Duloxetine — Administration of duloxetine
  Other Names: Cymbalta
  Arms: Control Arm

SUMMARY:
Chemotherapy induced peripheral neuropathy (CIPN) is a frequent and disabling complication of systemic chemotherapy, particularly with oxaliplatin or taxanes. The incidence of CIPN is variable but approximately 30-40% of patients treated with neurotoxic chemotherapy agents develop CIPN after long-term use of taxanes or oxaliplatin.

This CIPN is essentially a sensory peripheral neuropathy with pain manifested by unpleasant symptoms such as numbness, tingling, and less frequently shooting/burning pain. These symptoms spread proximally to affect both lower and upper extremities in a characteristic "stocking and glove" distribution.

Many symptoms of CIPN may resolve completely for some patients. However, CIPN is only partly reversible for most. In the worst instances, it does not appear to be reversible at all and can even increase over time.

CIPN is difficult to manage. Only duloxetine is recommended, based on the positive result of a randomized phase III double-blind placebo-controlled crossover trial. The use of duloxetine resulted in a greater reduction in pain and was effective in decreasing numbness and tingling in the feet. But, systemic antidepressants are often associated with toxicities and patients often refuse or abandon the treatment.

Capsaicin inhibits neural transmission in sensory axons and has been proven as effective on the intensity of pain for post-herpetic neuralgia and human immunodeficiency virus-associated neuropathy. Efficacy appears at one month and persists for at least 2 months.

Only a few studies focused on the efficacy of capsaicin 179 mg patch on the intensity of CIPN-induced pain. These non-randomized studies show that more than 50% of patients have a reduction in pain intensity of more than 30%.

Until now, no clinical trial has compared the efficacy of the capsaicin 179 mg patch with duloxetine.

Accordingly, this open-label phase 3, randomized, multicenter trial, will compare efficacy and safety of capsaicin patch with oral duloxetine on painful CIPN persisting more than 3 months after the end of the responsible chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patient with CIPN manifested by painful symptoms such as numbness and / or tingling and / or burning pain in fingers / hands and toes / feet with a typical distribution in "gloves and socks" beginning after neurotoxic chemotherapy
* Painful CIPN as expressed by the BPI-SF (average pain) as ≥ 4/10
* CIPN persisting at least 1 month after completion of chemotherapy with taxanes and/or platinum salts and sensory CIPN grade ≥ 2 according to the NCI Common Toxicity Criteria for Adverse Events (CTCAE v.5.0) grading scale
* Stable doses in the 4 weeks before screening, of concomitant neuropathic pain medication (antiepileptic drugs)
* Healthy and non-irritated skin on the areas to be treated
* Absence of neurotoxic chemotherapy planned during the next 6 months after inclusion
* Patient affiliated to a social security scheme
* > 18 years old
* Signed written informed consent form

Exclusion Criteria:

* Presence of known carcinomatous meningitis
* Pre-existing known peripheral neuropathy of another aetiology (alcohol, diabetes, …)
* Hypersensitivity to Capsaicin or contra-indications to duloxetine (e.g imatinib, tamoxifen)
* Patient already treated for this neuropathy with Capsaicin patches
* Patient treated by antidepressant drugs at time of inclusion
* Uncontrolled hypertension (systolic blood pressure ≥ 180 mmHg or diastolic blood pressure ≥ 90 mmHg) or recent history (<3 months) of cardiovascular events (stroke, heart attack, pulmonary embolism)
* Patients with known severe renal or hepatic failure
* Breastfeeding or pregnant women
* Persons deprived of liberty or guardianship (including curatorship)
* Patient unable to undergo regular medical follow-up for geographical, social or psychological.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 274 (Estimated)
Dates: Start 2023-10-20 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
The primary objective is to demonstrate that capsaicin 179 mg patch once compared to duloxetine daily, improves painful CIPN after a 5-week treatment period. | 5 weeks
  The primary endpoint will be the percentage of painful CIPN patients experiencing a 30% improvement in their average pain severity score at 6 weeks compared to baseline (measured on day 1 of week 6).
  Patient-reported pain severity will be quantified using the Brief Pain Inventory-Short Form (BPI-SF). The BPI-SF contains four items assessing average, worst, least, and immediate pain severity in the last 24 hours. Pain severity items are scored using an 11-point numeric rating scale (0 = no pain; 10 = pain as bad as you can imagine).
  In this study, we choose the "average" pain severity score as our primary outcome measure, following recommendations from the Initiative on Methods, Measurement, and Pain Assessment in Clinical Trials (IMMPACT).

CONTACTS AND LOCATIONS:
Overall Officials: François Xavier PILOQUET, MD, Study Director — Institut de Cancérologie de l'Ouest
Locations (11):
- France (11):
  - Institut de Cancérologie de l'Ouest, Angers
  - CHU Bordeaux, Bordeaux
  - Centre François Baclesse, Caen
  - CHU Grenoble, Grenoble
  - Polyclinique Chenieux, Limoges
  - Centre Léon Bérard, Lyon
  - "L'Hôpital Privé du Confluent ", Nantes
  - Centre Antoine Lacassagne, Nice
  - Institut de Cancérologie de l'Ouest, Saint-Herblain
  - Institut de Cancérologie Strasbourg Europe, Strasbourg
  - Institut Claudius Regaud -IUCT-O, Toulouse

IPD SHARING:
Plan to Share IPD: No